CLINICAL TRIAL: NCT03503643
Title: Cryoablation: An Observational Study of Hemi-Gland Cryoablation Outcomes for Prostate Cancer at University of California at Los Angeles (UCLA)
Brief Title: Hemi-Gland Cryoablation for Prostate Cancer at UCLA
Status: Enrolling by invitation | Type: Observational
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 17-001084
Record Dates: First submitted 2018-03-29; First posted 2018-04-20 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma; Prostate Disease
Keywords: prostate cancer; cryoablation
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Diseases | interventions — Cryotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Hemigland Cryoablation — Hemigland cryoablation for the treatment of prostate cancer
  Other Names: cryotherapy

SUMMARY:
This is a prospective data collection of men who are electing to undergo prostate hemi-gland cryoablation.

The purpose of this observational research study is to investigate the localized treatment of prostate cancer using hemi-gland cryoablation.

UCLA patients undergoing hemi-gland cryoablation are a unique cohort compared to prior research because all patients at UCLA have had a pre-treatment multi-parametric MRI and Ultrasound fusion targeted biopsy; they will be followed in a similar fashion. This results in more precise assessment of a target region of cancer for ablation which may, in turn, result in improved clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient has undergone or has elected to undergo hemi-gland cryoablation at UCLA
* Low or intermediate risk prostate cancer (Gleason ≤ 7) or select high-risk patients (Gleason 8 prostate cancer).
* Prostate volume of ≤ 70 cc
* Ability to complete informed consent form

Exclusion criteria:

* Medical contraindication to follow-up multi-parametric magnetic resonance imaging (mpMRI) or prostate biopsy
* Patients unable to tolerate general or regional anesthesia.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are candidates for hemi-gland cryoablation, and elect this treatment option as a standard of care procedure, will be considered for our clinical study and analysis of their outcomes. Subjects will provide informed consent to participate in this study during standard of care clinical visits at the Clark Urology Center at UCLA. Subjects will provide informed consent to allow study staff to abstract data from their medical records.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-09-14 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Response to Cancer Treatment | 6 months
  Our primary endpoint will be a patient's clinical response to cancer treatment, specifically, the degree of prostate cancer on a post-treatment fusion biopsy compared to pre-treatment.

SECONDARY OUTCOMES:
Quality of Life Assessment - Urinary Function | 6 months
  Comparison of urinary function pre- and post-treatment will be obtained using the International Prostate Symptom Score (IPSS) and the Expanded Prostate Cancer Index Composite (EPIC-26) questionnaires to report combined overall urinary function assessments.

OTHER OUTCOMES:
Quality of Life Assessment - Erectile Function | 6 months
  Comparison of erectile function pre- and post-treatment will be obtained using the 5-Item International Index of Erectile Function (IIEF-5) Sexual Health Inventory for Men and the Expanded Prostate Cancer Index Composite (EPIC-26) questionnaires to report combined overall erectile function assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard S Marks, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weiner AB, Proudfoot JA, Aker M, Cardenas M, Gonzalez S, Kelly E, Davicioni E, Sisk AE Jr, Brisbane WG, Marks LS. Genomic Biomarker for Prostate Cancer Focal Therapy: Post Hoc Assessment of a Phase II Clinical Trial. JCO Precis Oncol. 2025 Sep;9:e2500535. doi: 10.1200/PO-25-00535. Epub 2025 Sep 17. PMID 40961406